CLINICAL TRIAL: NCT00490724
Title: An Exploratory Study of JNS004 (Nesiritide) in Patients With Acute Heart Failure (J2)
Brief Title: An Exploratory Study of Nesiritide in Participants With Acute Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013903; JNS004-JPN-02
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-12

CONDITIONS: Heart Failure, Congestive
Keywords: Heart failure, congestive; Nesiritide and; JNS004
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nesiritide (1+0.01) (Experimental): Intravenous bolus treatment will be administered over 1 minute (min) at a dose of 1 microgram per kilogram (mcg/kg) followed by 24 hour intravenous infusion which is comprised of Period 1 (fixed-dose) with dose of 0.01 mcg/kg/min and Period 2 (flexible-dose) where dosage will be increased by 0.005 mcg/kg/min every 3 hours. Total dosage to be administered will be 15.4 to 35.2 mcg/kg.
  Interventions: Drug: Nesiritide (1+0.01)
- Nesiritide (2+0.005) (Experimental): Intravenous bolus treatment will be administered over 1 minute (min) at a dose of 2 microgram per kilogram (mcg/kg) followed by 24 hour intravenous infusion which is comprised of Period 1 (fixed-dose) with dose of 0.005 mcg/kg/min and Period 2 (flexible-dose) where dosage will be increased by 0.005 mcg/kg/min every 3 hours. Total dosage to be administered will be 9.2 to 31.7 mcg/kg.
  Interventions: Drug: Nesiritide (2+0.005)
- Nesiritide (2+0.01) (Experimental): Intravenous bolus treatment will be administered over 1 minute (min) at a dose of 2 microgram per kilogram (mcg/kg) followed by 24 hour intravenous infusion which is comprised of Period 1 (Fixed-dose) with dose of 0.01 mcg/kg/min and Period 2 (Flexible-dose) where dosage will be increased by 0.005 mcg/kg/min every 3 hours. Total dosage to be administered will be 16.4 to 36.2 mcg/kg.
  Interventions: Drug: Nesritide (2+0.01)

INTERVENTIONS:
Drug: Nesiritide (1+0.01) — Intravenous bolus treatment will be administered over 1 minute (min) at a dose of 1 microgram per kilogram (mcg/kg) followed by 24 hour intravenous infusion which is comprised of Period 1 (fixed-dose) with dose of 0.01 mcg/kg/min and Period 2 (flexible-dose) where dosage will be increased by 0.005 mcg/kg/min every 3 hours. Total dosage to be administered will be 15.4 to 35.2 mcg/kg.
  Arms: Nesiritide (1+0.01)
Drug: Nesiritide (2+0.005) — Intravenous bolus treatment will be administered over 1 minute (min) at a dose of 2 microgram per kilogram (mcg/kg) followed by 24 hour intravenous infusion which is comprised of Period 1 (fixed-dose) with dose of 0.005 mcg/kg/min and Period 2 (flexible-dose) where dosage will be increased by 0.005 mcg/kg/min every 3 hours. Total dosage to be administered will be 9.2 to 31.7 mcg/kg.
  Arms: Nesiritide (2+0.005)
Drug: Nesritide (2+0.01) — Intravenous bolus treatment will be administered over 1 minute (min) at a dose of 2 microgram per kilogram (mcg/kg) followed by 24 hour intravenous infusion which is comprised of Period 1 (Fixed-dose) with dose of 0.01 mcg/kg/min and Period 2 (Flexible-dose) where dosage will be increased by 0.005 mcg/kg/min every 3 hours. Total dosage to be administered will be 16.4 to 36.2 mcg/kg.
  Arms: Nesiritide (2+0.01)

SUMMARY:
The purpose of this exploratory study is to assess the efficacy and safety of nesiritide in participants with acute (a quick and severe form of illness in its early stage) heart failure (when the heart inadequately pumps blood through the body) including acute exacerbation of chronic (lasting a long time) heart failure, administered intravenous (into a vein) bolus (a large amount) followed by intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle).

DETAILED DESCRIPTION:
This is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), multi-center (when more than 1 hospital or medical school team work on a medical research study), randomized (study medication assigned by chance), stepwise, bolus plus intravenous infusion, fixed-flexible (arbitrary dose titration [slow increase in drug dosage, guided by participant's responses]) study. The study consists of 3 periods: Observation period (from the time of obtaining consent to the start of study treatment), Treatment period, and Follow-up period (from 24 hours after the initiation of study treatment [discontinuation] to 30 days after the initiation of study treatment). The participants will be randomly assigned to 1 of the following 3 treatment groups: 2+0.005 group, 1+0.01 group and 2+0.01 group. The treatment period consists of treatment with bolus injection (over 1 minute) followed by intravenous infusion (over 24 hours: Period 1 [fixed-dose period] of 3 hours and Period 2 [flexible-dose period] of 21 hours).The study will be conducted stepwise and hence, initially participants will be randomly assigned to 1 of the following 2 groups: 1+0.01 group and 2+0.005 group. Participants will receive nesiritide at an initial dose of 0.005 or 0.01 microgram per kilogram per minute (mcg/kg/min), and the dose escalation of 0.005 mcg/kg/min per dose will be conducted every 3 hours up to maximum of 0.03 mcg/kg/min in Period 2. Safety data of at least 5 participants will be assessed for each group, and after confirming the safety of 2 groups, the participants will be assigned to third group of nesiritide 2 microgram per kilogram (mcg/kg) +0.01 mcg/kg/min. Then participants will be followed up to a maximum of 30 days after the initiation of study treatment, in follow-up period. Participants will primarily be evaluated for the effect of nesiritide on hemodynamic parameters such as pulmonary capillary wedge pressure (PCWP), or if it is unmeasurable then it will be complemented with pulmonary arterial diastolic pressure (PADP). Participants' safety will also be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with acute heart failure (including acute exacerbation of chronic heart failure) requiring hospitalization whose placement of right-heart catheter (flexible, tube-like tool used to take fluids out or put fluids into the body) is judged to be possible and useful for treatment
* Participants with findings of pulmonary (having to do with the lungs) congestion on a chest X-ray (an image of a site produced on photographic film by X-rays passing through the site) film taken within 12 hours before starting the treatment
* Participants with 2 systolic blood pressure (SBP: refers to blood pressure [pressure of the blood on the arteries and other blood vessel] when the heart beats while pumping blood) values greater than or equal to 100 millimeters of mercury (mmHg) measured at an interval of at least 15 minutes in the hemodynamic (related to blood flow) assessment in observation period
* In a hemodynamic assessment in observation period, participants with 2 pulmonary capillary wedge pressure (PCWP [if it is not available, pulmonary arterial diastolic pressure {PADP}]) values greater than or equal to 18 mmHg measured at an interval of at least 15 minutes and the second measurement value is within positive 20 percent (%) and negative 20% compared with the first 1

Exclusion Criteria:

* Participants with severe (very serious, life threatening) hepatic (to do with liver) impairment or renal (to do with kidney) impairment, cancer (abnormal tissue that grows and spreads in the body until it kills), or malignant (cancerous) tumor (a mass in a specific area)
* Participants who are or may be pregnant or breast-feeding
* Participants receiving non-invasive (puncture, opening or cutting of the skin) positive pressure ventilation (NIPPV) or scheduled to receive this during the study period
* Participants who received treatment with another investigational product within 4 weeks before the initiation of investigational treatment or who were enrolled in a clinical study of nesiritide in the past
* Participants who received prohibited concomitant medications within 3 hours before the initiation of investigational treatment or those who are receiving such a medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (11):
- Japan (11):
  - Amagasaki
  - Chikushino-shi
  - Hiroshima
  - Ikoma
  - Komatsushima
  - Kumamoto
  - Moriyama
  - Osaka
  - Saitama
  - Tokyo
  - Yokohama

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 67 participants provided consent, out of these 61 participants were assigned to the study treatment.
Groups:
- Nesiritide (1+ 0.01): Intravenous bolus treatment was administered over 1 minute (min) at a dose of 1 microgram per kilogram (mcg/kg) followed by 24 hour intravenous infusion which was comprised of Period 1 (fixed-dose) with dose of 0.01 mcg/kg/min and Period 2 (flexible-dose) where dosage were increased by 0.005 mcg/kg/min every 3 hours. Total dosage administered was 15.4 to 35.2 mcg/kg.
- Nesiritide (2+0.005): Intravenous bolus treatment was administered over 1 minute (min) at a dose of 2 microgram per kilogram (mcg/kg) followed by 24 hour intravenous infusion which was comprised of Period 1 (Fixed-dose) with dose of 0.005 mcg/kg/min and Period 2 (Flexible-dose) where dosage were increased by 0.005 mcg/kg/min every 3 hours. Total dosage administered was 9.2 to 31.7 mcg/kg.
- Nesiritide (2+0.01): Intravenous bolus treatment was administered over 1 minute (min) at a dose of 2 microgram per kilogram (mcg/kg) followed by 24 hour intravenous infusion which was comprised of Period 1 (Fixed-dose) with dose of 0.01 mcg/kg/min and Period 2 (Flexible-dose) where dosage were increased by 0.005 mcg/kg/min every 3 hours. Total dosage administered was 16.4 to 36.2 mcg/kg.
Period: Period I
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Started | 21 | 20 | 20
Completed | 21 | 20 | 19
Not Completed | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Period: Period II
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Started | 21 | 20 | 19
Completed | 18 | 19 | 16
Not Completed | 3 | 1 | 3
Not completed — Treatment Discontinuation | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: The per protocol set (PPS) included all participants who met the principal criteria for eligibility, received at least 1 dose of study medication and had one efficacy assessment after randomization except those participants who had significant protocol deviations
Groups:
- Total: Total of all reporting groups
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01) | Total
Number analyzed (Participants) | 19 | 20 | 17 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were analysed for the per protocol set (PPS). The PPS included all participants who met the principal criteria for eligibility, received at least 1 dose of study medication and had 1 efficacy assessment after randomization except those participants who had significant protocol deviations.
  Years | 71.1 (14.1) | 67.5 (13.5) | 64.9 (11.6) | 67.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants] — The PPS included all participants who met the principal criteria for eligibility, received at least 1 dose of study medication and had 1 efficacy assessment after randomization except those participants who had significant protocol deviations.
  Participants
    Female | 8 | 6 | 7 | 21
    Male | 11 | 14 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Capillary Wedge Pressure (PCWP or Pulmonary Arterial Diastolic Pressure[PADP]) at 3 Hours
Description: Change in PCWP was unmeasurable, therefore it was complemented with PADP. PCWP was measured by pulmonary artery catheterization and provided an indirect measure of left atrial pressure.
Time Frame: Baseline and 3 Hours
Population: The per protocol set (PPS) included participants who met the eligibility criteria, received at least 1 dose of study medication and had one efficacy assessment after randomization except those who had significant protocol deviations.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Millimeters of Mercury (mmHg)
  Baseline | 27.7 (8.2) | 24.8 (6.3) | 29.7 (6.6)
  Change at 3 hours | -6.7 (5.8) | -5.4 (6.3) | -6.2 (6.8)

2. Secondary Outcome: Change From Baseline in Mean Right Atrial Pressure (MRAP) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 15 and 24 Hour
Description: The MRAP was a measured hemodynamic parameter. MRAP was measured using a Swan-Ganz catheter.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 15 and 24 Hour
Population: The PPS included participants who met the eligibility criteria, received at least 1 dose of study medication and had one efficacy assessment after randomization except those who had significant protocol deviations. Here, N=the participants evaluated for this measure and n=the participants evaluated for this measure at a particular time point.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 18 | 16
Millimeters of mercury
  Baseline (n=19,18,16) | 14.5 (9.0) | 10.3 (6.8) | 13.1 (6.2)
  Change at 0.25 hour (n=19,17,16) | -1.9 (3.4) | -2.5 (3.0) | -2.6 (2.4)
  Change at 0.5 hour (n=19,18,16) | -2.6 (4.0) | -3.1 (3.2) | -3.4 (2.7)
  Change at 1 hour (n=19,18,16) | -3.6 (3.5) | -2.7 (3.4) | 3.6 (3.4)
  Change at 1.5 hour (n=19,18,16) | -3.8 (6.3) | -3.4 (4.5) | -3.8 (3.3)
  Change at 2 hour (n=19,18,16) | -4.3 (6.2) | -2.8 (4.3) | -3.4 (3.8)
  Change at 2.5 hour(n=19,18,16) | -4.2 (4.7) | -2.5 (4.1) | -3.2 (4.9)
  Change at 3 hour (n=19,18,16) | -4.4 (5.5) | -2.5 (3.7) | -2.9 (4.7)
  Change at 4 hour (n=19,17,16) | -4.9 (4.8) | -2.0 (4.2) | -2.9 (6.0)
  Change at 5 hour (n=18,17,16) | -5.0 (5.1) | -3.0 (4.6) | -2.9 (7.1)
  Change at 6 hour (n=18,17,16) | -5.1 (4.8) | -3.3 (3.7) | -3.1 (6.9)
  Change at 12 hour (n=17,17,16) | -5.9 (6.7) | -3.4 (3.2) | -4.3 (4.2)
  Change at 15 hour (n=2,1,0) | 1.0 (2.8) | -3.5 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n=14,17,14) | -5.2 (4.6) | -4.5 (4.7) | -5.0 (5.3)

3. Secondary Outcome: Change From Baseline in Pulmonary Arterial Systolic Pressure (PASP) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Description: The PASP was a measured hemodynamic parameters. PASP was assessed by Swan-Ganz catheter.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Population: The PPS included participants who met the eligibility criteria, received at least 1 dose of study medication and had one efficacy assessment after randomization except those who had significant protocol deviations. Here, n=the participants evaluated for this measure at a particular time point.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Millimeters of mercury
  Baseline (n=19,20,17) | 55.9 (16.5) | 51.3 (11.1) | 59.8 (12.0)
  Change at 0.25 hour (n=19,19,17) | -3.6 (6.2) | -8.2 (7.9) | -4.2 (5.2)
  Change at 0.5 hour (n=19,20,17) | -5.3 (7.6) | -8.7 (9.5) | -5.5 (4.8)
  Change at 1 hour (n=19,20,17) | -7.0 (8.8) | -8.7 (9.5) | -7.4 (5.7)
  Change at 1.5 hour (n=19,20,17) | -6.2 (9.1) | -7.6 (8.0) | -8.8 (6.6)
  Change at 2 hour (n=19,20,17) | -7.2 (8.6) | -6.8 (9.1) | -7.0 (6.3)
  Change at 2.5 hour (n=19,20,17) | -7.0 (9.8) | -5.9 (7.4) | -6.6 (6.9)
  Change at 3 hour (n=19,20,17) | -9.4 (10.5) | -6.1 (8.9) | -6.4 (7.8)
  Change at 4 hour (n=19,19,17) | -10.2 (12.2) | -5.7 (9.2) | -7.5 (6.9)
  Change at 5 hour (n=18,19,17) | -10.0 (12.6) | -6.8 (9.5) | -8.2 (6.0)
  Change at 6 hour (n=18,19,17) | -9.9 (12.1) | -6.1 (9.7) | -10.1 (7.7)
  Change at 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 13.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 12 hour (n=17,19,17) | -11.3 (12.9) | -9.1 (10.4) | -12.7 (7.7)
  Change at 15 hour (n=2,1,0) | 6.0 (4.9) | 6.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n=14,19,15) | -9.3 (10.5) | -10.4 (11.9) | -12.2 (7.6)

4. Secondary Outcome: Change From Baseline in Pulmonary Arterial Diastolic Pressure (PADP) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Description: The PADP was a measured hemodynamic parameter. Normal range of PADP is 8 to 15 millimeters of mercury (mmHg). PADP was assessed by Swan-Ganz catheter.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Millimeters of mercury
  Baseline (n=19,20,17) | 26.5 (8.4) | 24.2 (7.4) | 30.1 (8.0)
  Change at 0.25 hour (n=19,19,17) | -1.6 (3.1) | -6.1 (4.6) | -4.6 (3.3)
  Change at 0.5 hour (n=19,20,17) | -2.8 (4.0) | -6.9 (5.6) | -6.6 (4.3)
  Change at 1 hour (n=19,20,17) | -4.0 (6.0) | -5.7 (6.1) | -7.0 (4.4)
  Change at 1.5 hour (n=19,20,17) | -3.2 (6.5) | -5.6 (5.5) | -6.9 (4.3)
  Change at 2 hour (n=19,20,17) | -4.6 (6.4) | -5.4 (5.3) | -5.6 (5.3)
  Change at 2.5 (n=19,20,17) | -3.5 (6.9) | -3.6 (4.8) | -6.2 (5.9)
  Change at 3 hour (n=19,20,17) | -4.7 (6.7) | -3.6 (5.3) | -5.9 (6.0)
  Change at 4 hour (n=19,19,17) | -6.7 (7.1) | -4.4 (5.6) | -6.5 (5.6)
  Change at 5 hour (n=18,19,17) | -6.3 (7.5) | -4.5 (5.4) | -6.5 (5.2)
  Change at 6 hour (n=18,19,17) | -6.7 (6.9) | -4.1 (5.6) | -8.0 (5.8)
  Change at 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 14.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 12 hour (n=17,19,17) | -6.8 (8.3) | -5.6 (5.2) | -8.9 (7.6)
  Change at 15 hour (n=2,1,0) | 3.5 (4.9) | 3.5 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n=14,19,15) | -5.7 (5.9) | -6.0 (6.4) | -8.0 (6.4)

5. Secondary Outcome: Change From Baseline in Mean Pulmonary Arterial Pressure (MPAP) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Description: The MPAP was a measured hemodynamic parameter. MPAP was measured using a Swan-Ganz catheter.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Millimeters of mercury
  Baseline (n=19,20,17) | 38.2 (10.8) | 34.5 (8.5) | 42.6 (7.8)
  Change at 0.25 hour (n=19,19,17) | -2.3 (3.8) | -7.0 (5.5) | -4.9 (4.6)
  Change at 0.5 hour (n=19,20,17) | -3.2 (5.0) | -7.6 (7.2) | -5.5 (4.4)
  Change at 1 hour (n=19,20,17) | -5.0 (5.9) | -6.7 (7.4) | -7.8 (5.4)
  Change at 1.5 hour (n=19,20,17) | -4.8 (7.4) | -6.7 (6.6) | -7.8 (5.8)
  Change at 2 hour (n=19,20,17) | -5.3 (7.0) | -5.7 (7.1) | -6.4 (5.8)
  Change at 2.5 hour (n=19,20,17) | -5.4 (7.0) | -4.9 (7.8) | -6.7 (6.5)
  Change at 3 hour (n=19,20,17) | -6.5 (7.6) | -5.6 (8.5) | -5.9 (6.1)
  Change at 4 hour (n=19,19,17) | -8.3 (8.3) | -5.0 (7.1) | -7.1 (6.1)
  Change at 5 hour (n=18,19,17) | -7.5 (8.7) | -6.3 (6.8) | -7.8 (4.7)
  Change at 6 hour (n=18,19,17) | -7.7 (8.4) | -6.0 (7.2) | -9.5 (7.0)
  Change at 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 12.5 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 12 hour (n=17,19,17) | -8.1 (10.6) | -7.8 (6.7) | -11.3 (7.0)
  Change at 15 hour (n=2,1,0) | 3.5 (7.1) | 4.5 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n=14,19,15) | -7.0 (7.2) | -8.6 (9.0) | -11.0 (6.1)

6. Secondary Outcome: Change From Baseline in Pulmonary Capillary Wedge Pressure (PCWP) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Description: The PCWP was a measured hemodynamic parameter. It was the blood pressure, recorded after wedging a catheter in a small pulmonary artery; believed to reflect the pressure in the pulmonary capillaries. It was measured by pulmonary artery catheterization and provided an indirect measure of left atrial pressure.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 14 | 18 | 12
Millimeters of mercury
  Baseline (n=14,18,14) | 27.0 (6.0) | 24.3 (5.1) | 30.2 (7.0)
  Change at 0.25 hour (n=14,17,13) | -3.5 (3.7) | -5.5 (3.9) | -5.1 (6.0)
  Change at 0.5 hour (n=14,18,13) | -5.1 (3.4) | -7.9 (5.5) | -7.5 (5.5)
  Change at 1 hour (n=14,18,12) | -5.6 (4.5) | -7.6 (5.3) | -8.5 (5.8)
  Change at 1.5 hour (n=14,18,12) | -5.5 (3.5) | -6.5 (4.7) | 9.0 (6.2)
  Change at 2 hour (n=14,18,12) | -5.1 (3.8) | -6.3 (5.1) | -7.6 (6.0)
  Change at 2.5 hour (n=14,18,12) | -5.6 (4.9) | -5.0 (5.7) | -7.9 (6.4)
  Change at 3 hour (n=14,18,12) | -6.5 (4.6) | -4.9 (6.2) | -7.9 (5.5)
  Change at 4 hour (n=14,17,12) | -7.9 (3.8) | -4.9 (6.2) | -7.5 (5.8)
  Change at 5 hour (n=12,17,12) | -8.6 (2.9) | -5.8 (5.8) | -8.0 (5.0)
  Change at 6 hour (n=12,17,12) | -9.5 (3.0) | -5.6 (4.9) | -11.2 (5.9)
  Change at 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 12.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 12 hour (n=10,17,12) | -9.9 (3.6) | -7.8 (4.9) | -11.8 (6.5)
  Change at 15 hour (n=1,1,0) | -4.5 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | -1.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n=9,17,10) | -9.7 (6.6) | -7.2 (5.5) | -10.5 (3.9)

7. Secondary Outcome: Change From Baseline in Cardiac Output (CO) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Description: The CO was a measured cardiopulmonary hemodynamic parameter. It is the volume of blood expelled by the ventricles of the heart with each beat. It was calculated as the product of stroke volume (output of either ventricle per heartbeat) and the number of beats per minute. Cardiac output is commonly measured by the thermodilution technique.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liter per minute
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Liter per minute
  Baseline (n=19,20,17) | 4.4026 (1.4463) | 3.9768 (1.2767) | 4.0971 (1.4259)
  Change at 0.25 hour (n=19,19,17) | 0.2947 (0.7227) | 0.5686 (0.7616) | 0.2912 (0.9378)
  Change at 0.5 hour (n=19,20,17) | 0.3721 (0.6143) | 0.8102 (0.9328) | 1.4147 (1.2028)
  Change at 1 hour (n=19,20,17) | 0.3668 (0.9398) | 0.7838 (0.7643) | 1.1382 (0.6744)
  Change at 1.5 hour (n=19,20,17) | 0.2795 (1.1145) | 0.5947 (1.1077) | 0.7206 (1.0939)
  Change at 2 hour (n=19,20,17) | 0.3026 (1.3596) | 0.3497 (1.0715) | 0.3500 (0.7163)
  Change at 2.5 hour (n=19,20,17) | -0.3105 (1.1770) | 0.0292 (0.6977) | 0.3029 (0.9547)
  Change at 3 hour (n=19,20,17) | 0.0095 (1.0695) | 0.1597 (0.7112) | -0.0265 (0.8170)
  Change at 4 hour (n=19,19,17) | -0.2742 (0.9836) | 0.1435 (0.7650) | 0.1912 (0.5167)
  Change at 5 hour (n=18,19,17) | -0.3356 (1.2717) | 0.1472 (0.6739) | 0.2676 (0.9761)
  Change at 6 hour (n=18,19,17) | -0.5706 (1.4351) | -0.1994 (0.6581) | 0.1735 (1.0341)
  Change at 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 0.3500 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 12 hour (n=16,19,17) | -0.5453 (0.8935) | -0.3177 (0.6534) | 0.2853 (1.2070)
  Change at 15 hour (n=2,1,0) | -0.4500 (0.5657) | 0.3000 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n=14,19,15) | -0.1246 (1.1352) | -0.3108 (0.8702) | -0.3200 (1.1894)

8. Secondary Outcome: Change From Baseline in Mean Blood Pressure (MBP) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15, 18, 21 and 24 Hour
Description: The MBP was a calculated hemodynamic parameter and the calculation was done on the basis of the measured hemodynamic parameters. MBP was calculated as sum of diastolic blood pressure (DBP) and (0.33*[SBP-DBP])
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15, 18, 21 and 24 Hour
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Millimeters of mercury
  Baseline (n=19,20,17) | 109.397 (15.868) | 106.169 (20.438) | 105.006 (17.781)
  Change at 0.25 hour (n=19,19,17) | -6.053 (6.452) | -9.167 (8.975) | -7.098 (14.093)
  Change at 0.5 hour (n=19,20,17) | -4.626 (7.316) | -9.930 (8.124) | -9.450 (10.543)
  Change at 1 hour (n=19,20,17) | -6.900 (8.890) | -7.863 (8.599) | -7.685 (12.821)
  Change at 1.5 hour (n=19,20,17) | -7.412 (12.835) | -10.181 (9.339) | 4.969 (11.997)
  Change at 2 hour (n=19,20,17) | -10.032 (11.474) | -11.149 (10.411) | -6.669 (9.468)
  Change at 2.5 hour (n=19,20,17) | -8.497 (14.396) | -12.516 (9.011) | -6.890 (10.768)
  Change at 3 hour (n=19,20,17) | -8.773 (14.660) | -11.666 (9.572) | -9.517 (11.114)
  Change at 4 hour (n=19,20,17) | -10.310 (12.873) | -10.858 (10.196) | -5.681 (11.438)
  Change at 5 hour (n=18,20,17) | -12.541 (11.645) | -9.301 (10.935) | -8.254 (11.070)
  Change at 6 hour (n=19,20,17) | -15.167 (17.875) | -12.241 (16.070) | -9.281 (12.960)
  Change at 9 hour (n=19,20,17) | -17.689 (17.866) | -9.287 (17.532) | -14.619 (14.311)
  Change at 12 hour (n=19,20,17) | -16.107 (19.174) | -13.113 (13.733) | -16.103 (15.392)
  Change at 15 hour (n=19,20,17) | -16.050 (18.244) | -11.584 (15.233) | -15.590 (13.885)
  Change at 18 hour (n=19,20,17) | -16.040 (21.176) | -16.331 (16.193) | -15.962 (16.456)
  Change at 21 hour (n=19,20,17) | -16.933 (18.362) | -14.267 (16.993) | -18.684 (20.086)
  Change at 24 hour (n= 19,20,16) | -16.590 (19.882) | -12.162 (17.803) | -11.135 (12.593)

9. Secondary Outcome: Change From Baseline in Cardiac Index (CI) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Description: The CI was a calculated hemodynamic parameter and the calculation was done on the basis of the measured hemodynamic parameters. CI was calculated by dividing CO and body surface area.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liter per minute per meter^2 (l/min/m^2)
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Liter per minute per meter^2 (l/min/m^2)
  Baseline (n=19,20,17) | 2.712 (0.826) | 2.356 (0.527) | 2.382 (0.549)
  Change at 0.25 hour (n=19,19,17) | 0.199 (0.442) | 0.305 (0.395) | 0.232 (0.540)
  Change at 0.5 hour (n=19,20,17) | 0.239 (0.357) | 0.443 (0.451) | 0.861 (0.783)
  Change at 1 hour (n=19,20,17) | 0.226 (0.555) | 0.445 (0.404) | 0.695 (0.443)
  Change at 1.5 hour (n=19,20,17) | 0.166 (0.673) | 0.293 (0.477) | 0.439 (0.603)
  Change at 2 hour (n=19,20,17) | 0.143 (0.758) | 0.165 (0.535) | 0.216 (0.459)
  Change at 2.5 hour (n=19,20,17) | -0.175 (0.672) | 0.042 (0.425) | 0.158 (0.492)
  Change at 3 hour (n=19,20,17) | -0.011 (0.613) | 0.092 (0.388) | 0.029 (0.560)
  Change at 4 hour (n=19,19,17) | -0.153 (0.556) | 0.055 (0.431) | 0.131 (0.324)
  Change at 5 hour (n=18,19,17) | -0.212 (0.733) | 0.061 (0.329) | 0.153 (0.572)
  Change at 6 hour (n=18,19,17) | -0.307 (0.732) | -0.127 (0.368) | 0.103 (0.622)
  Change at 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 0.185 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 12 hour (n=16,19,17) | -0.318 (0.518) | -0.201 (0.370) | 0.185 (0.780)
  Change at 15 hour (n=2,1,0) | -0.274 (0.331) | 0.186 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n= 14,19,15) | 0.054 (0.617) | -0.199 (0.507) | 0.148 (0.754)

10. Secondary Outcome: Change From Baseline in Stroke Volume (SV) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Description: The SV was a calculated hemodynamic parameter and the calculation was done on the basis of the measured hemodynamic parameters. Stroke volume is the volume of blood ejected from a ventricle at each beat of the heart, equal to the difference between the end-diastolic volume and the end-systolic volume. SV was calculated by dividing CO and heart rate (HR).
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter (ml)
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 17 | 19 | 17
milliliter (ml)
  Baseline (n=17,19,17) | 48.368 (18.272) | 49.126 (22.030) | 41.545 (12.290)
  Change at 0.25 hour (n=17,19,17) | 4.122 (9.604) | 3.305 (7.556) | 3.517 (8.589)
  Change at 0.5 hour (n=17,19,17) | 6.348 (8.940) | 6.887 (11.497) | 15.121 (13.429)
  Change at 1 hour (n=17,19,17) | 6.295 (9.587) | 8.442 (8.368) | 13.039 (7.426)
  Change at 1.5 hour (n=17,19,17) | 4.666 (11.659) | 7.722 (12.452) | 8.293 (9.497)
  Change at 2 hour (n=17,19,17) | 6.003 (14.727) | 6.877 (15.550) | 6.119 (8.270)
  Change at 2.5 hour (n=17,19,17) | 0.133 (12.357) | 1.768 (11.073) | 5.490 (9.857)
  Change at 3 hour (n=17,19,17) | 4.744 (12.370) | 2.865 (8.973) | 2.909 (8.238)
  Change at 4 hour (n=17,18,17) | 1.477 (10.205) | 2.888 (9.530) | 5.053 (5.633)
  Change at 5 hour (n=16,18,17) | 0.909 (16.362) | 4.339 (8.641) | 6.802 (9.925)
  Change at 6 hour (n=16,18,17) | -0.391 (15.734) | 2.685 (13.448) | 5.544 (9.810)
  Change at 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 8.792 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 12 hour (n=15,18,17) | 1.254 (13.051) | -1.357 (12.043) | 9.123 (12.779)
  Change at 15 hour (n=2,1,0) | -5.022 (1.839) | -0.955 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n=13,18,15) | 2.333 (16.239) | -1.421 (14.266) | 0.448 (11.288)

11. Secondary Outcome: Change From Baseline in Stroke Volume Index (SVI) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Description: The SVI was a calculated hemodynamic parameter and the calculation was done on the basis of the measured hemodynamic parameters. Stroke volume is the volume of blood ejected from a ventricle at each beat of the heart, equal to the difference between the end-diastolic volume and the end-systolic volume. The stroke volume index is a method of relating the stroke volume to the size of the person by dividing the stroke volume by the body surface area (BSA).
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter per meter^2
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 17 | 19 | 17
milliliter per meter^2
  Baseline (n=17,19,17) | 29.683 (11.141) | 28.655 (9.810) | 24.483 (6.016)
  Change at 0.25 hour (n=17,18,17) | 2.888 (5.948) | 1.853 (4.525) | 2.584 (5.200)
  Change at 0.5 hour (n=17,19,17) | 4.116 (5.692) | 3.775 (6.143) | 9.191 (8.552)
  Change at 1 hour (n=17,19,17) | 3.904 (5.927) | 4.892 (4.766) | 8.007 (4.936)
  Change at 1.5 hour (n=17,19,17) | 2.822 (7.127) | 3.900 (5.161) | 4.948 (5.142)
  Change at 2 hour (n=17,19,17) | 3.196 (7.954) | 3.526 (7.903) | 3.760 (5.210)
  Change at 2.5 hour n=17,19,17) | 0.394 (7.126) | 1.501 (6.587) | 3.052 (5.474)
  Change at 3 hour (n=17,19,17) | 2.751 (6.960) | 1.781 (5.369) | 2.091 (5.535)
  Change at 4 hour (n=17,18,17) | 1.097 (5.952) | 1.494 (5.568) | 3.142 (3.461)
  Change at 5 hour (n=16,18,17) | 0.525 (9.552) | 2.427 (4.530) | 4.146 (6.125)
  Change at 6 hour (n=16,18,17) | 0.320 (8.458) | 1.421 (7.082) | 3.319 (6.079)
  Change at 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 4.657 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 12 hour (n=15,18,17) | 1.100 (8.143) | -0.912 (6.992) | 5.610 (8.298)
  Change at 15 hour (n=2,1,0) | -3.357 (0.593) | -0.592 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n=13,18,15) | 1.690 (9.763) | -0.808 (7.217) | 0.590 (6.884)

12. Secondary Outcome: Change From Baseline in Systemic Vascular Resistance (SVR) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12 and 24 Hour
Description: The SVR was a calculated hemodynamic parameter and the calculation was done on the basis of the measured hemodynamic parameters. SVR was calculated by dividing (80*[MBP-MRAP]) and CO.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12 and 24 Hour
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dyne*second per centimeter^5
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 18 | 16
dyne*second per centimeter^5
  Baseline (n=19,18,16) | 1935.318 (687.715) | 2170.633 (896.353) | 2062.369 (894.394)
  Change at 0.25 hour (n=19,17,16) | -261.453 (301.208) | -366.981 (340.678) | -384.379 (651.980)
  Change at 0.5 hour (n=19,18,16) | -229.968 (250.083) | -453.601 (505.637) | -686.497 (784.338)
  Change at 1 hour (n=19,18,16) | -265.611 (419.843) | -456.113 (496.625) | -611.673 (640.704)
  Change at 1.5 hour (n=19,18,16) | -170.120 (551.743) | -328.746 (299.522) | -370.457 (458.264)
  Change at 2 hour (n=19,18,16) | -121.127 (652.720) | -308.987 (378.774) | -316.466 (580.484)
  Change at 2.5 hour (n=19,18,16) | 49.262 (797.660) | -292.112 (422.397) | -220.959 (357.619)
  Change at 3 hour (n=19,18,16) | -81.183 (487.205) | -297.880 (375.627) | -219.786 (545.724)
  Change at 4 hour (n=19,17,16) | -18.367 (467.058) | -339.457 (663.324) | -184.293 (396.692)
  Change at 5 hour (n=18,17,16) | 40.462 (592.227) | -254.269 (425.412) | -211.770 (375.316)
  Change at 6 hour (n=18,17,16) | 0.026 (562.942) | -68.635 (508.949) | -189.116 (493.764)
  Change at 12 hour (n=16,17,16) | 157.757 (743.728) | -26.925 (513.032) | -327.763 (648.264)
  Change at 24 hour (n=14,17,14) | -88.612 (390.796) | 68.641 (921.094) | -56.456 (477.960)

13. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Description: The PVR (force that opposes the flow of blood through a vascular bed) was a calculated hemodynamic parameter and the calculation was done on the basis of the measured hemodynamic parameters. PVR was calculated by dividing (80*[MPAP-PCWP]) and CO.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 15 and 24 Hour
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dyne*second/centimeter^5
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 14 | 18 | 14
dyne*second/centimeter^5
  Baseline (n=14,18,14) | 215.736 (124.776) | 208.714 (166.213) | 239.383 (122.453)
  Change at 0.25 hour (n=14,17,13) | -19.361 (79.932) | -40.647 (97.780) | -12.482 (86.016)
  Change at 0.5 hour (n=14,18,13) | -12.954 (70.125) | -23.263 (141.171) | -34.144 (100.492)
  Change at 1 hour (n=14,18,12) | -0.991 (93.305) | 1.964 (110.283) | -44.337 (116.971)
  Change at 1.5 hour (n=14,18,12) | 19.161 (57.701) | -2.975 (93.034) | -34.079 (109.876)
  Change at 2 hour (n=14,18,12) | 11.083 (69.935) | 23.400 (116.715) | -2.991 (104.337)
  Change at 2.5 hour (n=14,18,12) | 32.991 (59.277) | 11.609 (106.732) | 1.610 (107.365)
  Change at 3 hour (n=14,18,12) | 6.691 (88.625) | -2.667 (122.330) | 11.381 (109.961)
  Change at 4 hour (n=14,17,12) | 12.217 (103.059) | 3.797 (128.528) | -30.437 (89.235)
  Change at 5 hour (n=12,17,12) | 30.161 (73.755) | -10.958 (87.255) | -21.678 (97.090)
  Change at 6 hour (n=12,17,12) | 50.780 (117.927) | 10.104 (94.079) | -4.627 (107.473)
  Change at 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 2.017 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 12 hour (n=10,17,12) | 42.717 (116.928) | 20.625 (109.345) | -18.302 (132.041)
  Change at 15 hour (n=1,1,0) | 46.681 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | 116.667 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  Change at 24 hour (n=9,17,10) | 32.656 (76.762) | -29.072 (133.105) | -37.891 (137.587)

14. Secondary Outcome: Number of Participants With Dyspnea Symptoms Assessed by Borg Scale Score
Description: Assessment of Dyspnea (difficult or labored breathing) was done using Borg scale. It is a 10-point scale where following scores stands for severity of dyspnea: 0=no breathlessness at all; 0.5=very very slight (just noticeable); 1=very slight; 2=slight; 3=moderate; 4=somewhat severe; 5=severe; 7=very severe breathlessness; 9=very very severe (almost maximum) and 10=maximum.
Time Frame: Baseline, 1 h and 24 h
Population: The PPS included participants who met the eligibility criteria, received at least 1 dose of study medication and had one efficacy assessment after randomization except those who had significant protocol deviations. Here, N=the participants evaluated for this measure.
Measure: Number; unit: Participants
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 17 | 20 | 17
Participants
  Baseline:Score 0; at 1 hour:Score 0 | 1 | 2 | 4
  Baseline:Score 0.5; at 1 hour:Score 1 | 0 | 1 | 0
  Baseline:Score 1; at 1 hour:Score 0 | 1 | 1 | 0
  Baseline:Score 1; at 1 hour:Score 1 | 0 | 1 | 0
  Baseline:Score 1; at 1 hour:Score 2 | 0 | 2 | 0
  Baseline:Score 2; at 1 hour:Score 0 | 0 | 1 | 0
  Baseline:Score 2; at 1 hour:Score 0.5 | 0 | 1 | 1
  Baseline:Score 2; at 1 hour:Score 1 | 1 | 1 | 0
  Baseline:Score 2; at 1 hour:Score 2 | 2 | 0 | 2
  Baseline:Score 3; at 1 hour:Score 1 | 0 | 1 | 1
  Baseline:Score 3; at 1 hour:Score 2 | 2 | 2 | 3
  Baseline:Score 3; at 1 hour:Score 3 | 1 | 0 | 2
  Baseline:Score 4; at 1 hour:Score 3 | 1 | 1 | 1
  Baseline:Score 4; at 1 hour:Score 4 | 1 | 1 | 0
  Baseline:Score 5; at 1 hour:Score 3 | 0 | 0 | 1
  Baseline:Score 5; at 1 hour:Score 4 | 0 | 1 | 0
  Baseline:Score 5; at 1 hour:Score 5 | 0 | 1 | 0
  Baseline:Score 6; at 1 hour:Score 1 | 0 | 1 | 0
  Baseline:Score 6; at 1 hour:Score 3 | 0 | 0 | 1
  Baseline:Score 7; at 1 hour:Score 0 | 0 | 0 | 1
  Baseline:Score 7; at 1 hour:Score 2 | 1 | 0 | 0
  Baseline:Score 7; at 1 hour:Score 3 | 1 | 1 | 0
  Baseline:Score 7; at 1 hour:Score 7 | 1 | 0 | 0
  Baseline:Score 8; at 1 hour:Score 3 | 2 | 0 | 0
  Baseline:Score 9; at 1 hour:Score 3 | 1 | 0 | 0
  Baseline:Score 9; at 1 hour:Score 4 | 1 | 0 | 0
  Baseline:Score 10; at 1 hour:Score 4 | 0 | 1 | 0
  Baseline:Score 0; at 24 hour:Score 0 | 1 | 2 | 2
  Baseline:Score 0; at 24 hour:Score 1 | 0 | 0 | 0
  Baseline:Score 0.5; at 24 hour:Score 1 | 0 | 1 | 0
  Baseline:Score 1; at 24 hour:Score 0 | 1 | 1 | 0
  Baseline:Score 1; at 24 hour:Score 1 | 0 | 3 | 0
  Baseline:Score 2; at 24 hour:Score 0 | 0 | 1 | 0
  Baseline:Score 2; at 24 hour:Score 0.5 | 1 | 0 | 1
  Baseline:Score 2; at 24 hour:Score 1 | 0 | 1 | 1
  Baseline:Score 2; at 24 hour:Score 2 | 1 | 1 | 1
  Baseline:Score 3; at 24 hour:Score 0 | 1 | 0 | 3
  Baseline:Score 3; at 24 hour:Score 0.5 | 1 | 0 | 2
  Baseline:Score 3; at 24 hour:Score 1 | 2 | 1 | 1
  Baseline:Score 3; at 24 hour:Score 2 | 0 | 1 | 0
  Baseline:Score 4; at 24 hour:Score 0 | 1 | 0 | 0
  Baseline:Score 4; at 24 hour:Score 0.5 | 0 | 1 | 0
  Baseline:Score 4; at 24 hour:Score 1 | 0 | 1 | 0
  Baseline:Score 4; at 24 hour:Score 3 | 0 | 0 | 1
  Baseline:Score 5; at 24 hour:Score 0 | 0 | 1 | 0
  Baseline:Score 5; at 24 hour:Score 1 | 0 | 0 | 1
  Baseline:Score 5; at 24 hour:Score 2 | 0 | 1 | 0
  Baseline:Score 6; at 24 hour:Score 0 | 0 | 1 | 0
  Baseline:Score 6; at 24 hour:Score 3 | 0 | 0 | 1
  Baseline:Score 7; at 24 hour:Score 0 | 0 | 1 | 0
  Baseline:Score 7; at 24 hour:Score 1 | 1 | 0 | 0
  Baseline:Score 7; at 24 hour:Score 3 | 1 | 0 | 0
  Baseline:Score 7; at 24 hour:Score 4 | 0 | 0 | 1
  Baseline:Score 8; at 24 hour:Score 1 | 2 | 0 | 0

15. Secondary Outcome: Number of Participants With Dyspnea Symptoms Assessed by Likert Scale Score
Description: Assessment of Dyspnea was done using Likert scale. It is a 7-point scale where following scores stands for severity of dyspnea: 1=markedly better; 2=moderately better; 3=minimally better; 4=no change; 5=minimally worse; 6=moderately worse and 7= markedly worse
Time Frame: 3, 6 and 24 hour
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 13 | 15 | 17
Participants
  At 3 hour: Score 1 | 5 | 4 | 6
  At 3 hour: Score 2 | 2 | 4 | 2
  At 3 hour: Score 3 | 3 | 3 | 3
  At 3 hour: Score 4 | 3 | 4 | 5
  At 3 hour: Score 5 | 0 | 0 | 1
  At 6 hour: Score 1 | 6 | 6 | 4
  At 6 hour: Score 2 | 3 | 2 | 5
  At 6 hour: Score 3 | 1 | 4 | 5
  At 6 hour: Score 4 | 2 | 2 | 3
  At 24 hour: Score 1 | 4 | 7 | 8
  At 24 hour: Score 2 | 3 | 4 | 0
  At 24 hour: Score 3 | 1 | 1 | 4
  At 24 hour: Score 4 | 2 | 2 | 3

16. Secondary Outcome: Number of Participants With Orthopnea
Description: Assessment of dyspnea was done by measuring percentage of participants showing presence or absence of orthopnea (it is the sensation of breathlessness in the recumbent position, relieved by sitting or standing) symptoms
Time Frame: Baseline, 1 and 24 hour
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 18 | 20 | 17
Participants
  Baseline: 'Yes'; at 1 hour 'Yes' | 6 | 4 | 4
  Baseline: 'Yes'; at 1 hour 'No' | 7 | 7 | 1
  Baseline: 'No'; at 1 hour 'No' | 5 | 9 | 12
  Baseline: 'Yes'; at 24 hour 'Yes' | 1 | 2 | 1
  Baseline: 'Yes'; at 24 hour 'No' | 7 | 8 | 4
  Baseline: 'No'; at 24 hour 'No' | 6 | 9 | 10

17. Secondary Outcome: Number of Participants With Oxygen Therapy
Description: Assessment of dyspnea was done by measuring number of participants showing presence or absence of oxygen therapy.
Time Frame: Baseline,1 and 24 hour
Population: The PPS were the residual participants having a significant protocol deviation influencing the efficacy assessment, obtained by subtracting from the FAS population. Here, N=the participants evaluated for this measure and n=the participants evaluated for this measure at a particular time point.
Measure: Number; unit: Participants
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 18 | 20 | 17
Participants
  Baseline: 'Yes';at 1 hour 'Yes'(n=18,20,17 | 16 | 20 | 17
  Baseline: 'No';at 1 hour 'No'(n=18,20,17) | 2 | 0 | 0
  Baseline: 'Yes';at 24 hour 'Yes'(n=14,19,15) | 12 | 19 | 15
  Baseline:'No';at 24 hour 'No'(n=14,19,15) | 2 | 0 | 0

18. Secondary Outcome: Assessment of Dyspnea Using Percutaneous Arterial Oxygen Saturation (SpO2)
Description: Assessment of dyspnea was done by measuring SpO2 via pulse oximetry, by making the participant lye quietly in the post anesthesia care unit (PACU) and breathing room air (RA)
Time Frame: Baseline, 1, 2, 3, 6, 9, 12, 15 and 24 hour
Population: The PPS were the residual participants having a significant protocol deviation influencing the efficacy assessment, obtained by subtracting from the FAS population. Here,n=the participants evaluated for this measure at a particular time point.
Measure: Mean (Standard Deviation); unit: Percentage of SpO2
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Percentage of SpO2
  Baseline (n=19,20,17) | 96.5 (2.9) | 96.4 (2.3) | 96.9 (2.0)
  At 1 hour (n=18,20,17) | 96.6 (2.2) | 96.6 (2.2) | 96.4 (5.2)
  At 2 hour (n=19,20,17) | 96.8 (2.3) | 96.8 (2.4) | 97.7 (1.4)
  At 3 hour (n=19,20,17) | 96.7 (2.7) | 96.9 (2.6) | 98.4 (0.9)
  At 6 hour (n=13,15,17) | 97.6 (1.8) | 97.3 (1.9) | 97.5 (1.5)
  At 9 hour (n=0,1,0) | NA (NA) — No participant was analyzed for this time point | 100.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  At 15 hour (n=2,1,0) | 94.5 (3.5) | 99.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  At 24 hour (n=14,19,15) | 97.1 (1.8) | 97.1 (1.8) | 98.1 (1.8)

19. Secondary Outcome: Assessment of Dyspnea Using Respiratory Rate
Description: Assessment of dyspnea was done by measuring respiratory rate which is the number of times an organism breathes with the lungs (respiration) per unit time, usually per minute
Time Frame: Baseline, 1, 2, 3, 6, 9, 15 and 24 hour
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Breaths Per Minute (BrPM)
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Breaths Per Minute (BrPM)
  Baseline (n= 19,20,17) | 24.7 (7.8) | 25.6 (6.5) | 23.8 (7.8)
  At 1 hour (n= 18,20,17) | 24.0 (8.3) | 23.0 (3.9) | 22.6 (6.5)
  At 2 hour (n= 19,20,17) | 23.2 (7.7) | 22.1 (4.1) | 21.2 (6.2)
  At 3 hour (n= 19,20,17) | 22.7 (7.1) | 22.9 (5.1) | 20.4 (6.7)
  At 6 hour (n= 13,15,17) | 21.2 (3.7) | 21.8 (4.9) | 20.5 (4.9)
  At 9 hour (n= 0,1,0) | NA (NA) — No participant was analyzed for this time point | 22.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  At 15 hour (n=2,1,0) | 22.0 (7.1) | 33.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | NA (NA) — No participant was analyzed for this time point
  At 24 hour (n= 14,18,17) | 19.4 (3.9) | 20.8 (5.0) | 21.4 (4.3)

20. Secondary Outcome: Urinary Volume
Description: The urinary volume was measured because nesiritide has a diuretic effect. Measurement of hour urine was done in the observation period and treatment period. 1-hour urine before treatment initiation was measured in the observation period. In the treatment period, 1-hour urine for period 1 and 3-hour urine for period 2 was measured. Urinary volume was recorded for participants without urethral catheterization having spontaneous micturition when needed.
Time Frame: Baseline, 3 and 24 hour
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millliter
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Number analyzed (Participants) | 19 | 20 | 17
Millliter
  Baseline (n=15,19,15) | 83.9 (69.5) | 67.0 (36.1) | 79.7 (110.6)
  At 3 hour (n=19,20,17) | 539.9 (333.5) | 423.6 (289.4) | 545.1 (643.6)
  At 24 hour (n=19,20,17) | 1976.3 (1296.0) | 2296.9 (1278.7) | 2233.6 (1569.6)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days
Arm/Group | Nesiritide (1+ 0.01) | Nesiritide (2+0.005) | Nesiritide (2+0.01)
Serious Adverse Events (participants affected / at risk) | 3/21 | 3/20 | 4/19
Other Adverse Events (participants affected / at risk) | 18/21 | 16/20 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nesiritide (1+ 0.01) (N=21) | Nesiritide (2+0.005) (N=20) | Nesiritide (2+0.01) (N=19)
Cardiac failure (Cardiac disorders) | 1 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Cerebral infarction (Vascular disorders) | 0 | 1 | 0
Cerebral artery embolism (Vascular disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nesiritide (1+ 0.01) (N=21) | Nesiritide (2+0.005) (N=20) | Nesiritide (2+0.01) (N=19)
Infection (Infections and infestations) | 0 | 0 | 2
Cystitis (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 2 | 1
Delirium (Psychiatric disorders) | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0
Cholinergic syndrome (Nervous system disorders) | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 2 | 3 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 1 | 2
Peripheral circulatory failure (Vascular disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Glossoptosis (Gastrointestinal disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 3 | 2
Hepatic congestion (Hepatobiliary disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Catheter site pain (General disorders) | 1 | 0 | 0
Infusion site phlebitis (General disorders) | 1 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 2 | 2 | 2
Blood urine present (Investigations) | 2 | 1 | 2
Blood urea increased (Investigations) | 1 | 3 | 0
Blood potassium increased (Investigations) | 0 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 2 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 1
Basophil count increased (Investigations) | 0 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Laboratory test abnormal (Investigations) | 1 | 0 | 0
Protein total decreased (Investigations) | 1 | 0 | 0
Pulmonary arterial wedge pressure increased (Investigations) | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 1
Protein urine present (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the Sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the Sponsor requires.